CLINICAL TRIAL: NCT04240665
Title: Compensation Training to Improve Everyday Functioning of Older Adults With Mild Cognitive Impairment and Subjective Cognitive Complaints: The Digital Memory Notebook
Brief Title: The Digital Memory Notebook
Acronym: DMN
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1454000
Record Dates: First submitted 2019-11-10; First posted 2020-01-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Prodromal Alzheimer's Disease; Mild Cognitive Impairment; Subjective Cognitive Complaints
MeSH Terms: conditions — Cognitive Dysfunction | interventions — desmuslin

STUDY DESIGN:
Intervention Model Description: All participants will complete a curriculum involving 2-hour weekly sessions for 6-weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DMN Intervention (Experimental): Subjects will attend 2-hour weekly sessions for 6- weeks. Participants will continue to use the DMN application for 4-weeks after the intervention is complete.
  Interventions: Behavioral: Digital Memory Notebook (DMN) Application

INTERVENTIONS:
Behavioral: Digital Memory Notebook (DMN) Application — Subjects will be taught to utilize the DMN application through 2-hour weekly sessions for 6-weeks.

SUMMARY:
Compensatory aids (e.g., alarms, calendars) play an important supporting role when completing everyday tasks (e.g., appointments, medication management), and there is a growing body of scientific work suggesting that compensatory training improves daily functioning. However, traditional paper-based calendars and to-do-lists have limitations related to accumulation of information, difficulty retrieving information, and remembering to complete activities. Such limitations may be overcome using a digital format through organized digital files, search functions, and alarms. This pilot project proposes to train older adults at risk for cognitive decline to use the Digital Memory Notebook (DMN), a tablet-based application (app), to support everyday functioning. The primary goal is to obtain preliminary evidence that a 6-week, individual and group-based DMN training intervention results in demonstrable changes in target behaviors (e.g., goal-directed DMN use to support everyday activities) among older adults with mild cognitive impairment (MCI) and subjective cognitive complaints (SCC). Participants will complete a curriculum involving 2-hour weekly sessions for 6-weeks. Each week will cover a specific function of the DMN and will include standardized goal-setting and weekly homework targets. Following the 6-week intervention, participants will continue to use the DMN app for 4-weeks to evaluate stability. Participants will complete a questionnaire packet 1 week prior to the 6-week intervention, 1 week after the 6-week intervention, and 5 weeks following the 6-week intervention. MCI and SCC participants will complete separate 6-week individual or group interventions spaced two months apart at UCD.

DETAILED DESCRIPTION:
The manualized curriculum will involve 2-hour weekly sessions for 6-weeks. The study personnel will administer all intervention sessions. Each week will cover a specific function of the Digital Memory Notebook (DMN) and will include standardized goal-setting and weekly homework targets. A research assistant will assess homework adherence using a standardized form and through data extracted from the DMN (e.g., number of alarms set). Mild cognitive impairment (MCI) and subjective cognitive complaints (SCC) participants will complete separate 6-week individual or group interventions. Following the 6-week intervention, participants will continue to use the DMN app for 4-weeks to evaluate stability.

Participants will also be asked to complete questions about their medical background including history of traumatic brain injury or stroke, as well as any current medical conditions and questions regarding demographics including age, ethnicity, and education.

Potential participants will be told that participating in the study will involve completing questionnaires at 3 different time points within 12 weeks (i.e.,week 1, week 8, week 12), identifying a knowledgeable informant who will also complete questionnaires, participating in a 6-week course to learn how to use the DMN and to support everyday functioning, and to continue to use the DMN for one month following the intervention.

Information collected will be in the form of counts (e.g., number of alarms set) and number of minutes spent on the device. Specific content entered into the DMN will not be reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of subjective cognitive complaints (SCC) or Mild Cognitive Impairment (MCI)
* Adults at least 60 years of age (no upper age limit)
* Fluent in English
* Available informant (study partner) to complete surveys

Exclusion Criteria:

* Unable to consent
* Pregnant women
* Prisoners

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-11-11 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Real-time data extracted from the DMN Application | Change in number of entries assessed weekly from first weekly session through Week 6 weekly session and for 4 weeks after the completion of the last session
  data that is automatically collected by DMN (Calendar entries, to-do list entries, alarms set, journal entries)

SECONDARY OUTCOMES:
Participant Questionnaire Outcomes | Week 1, Week 8, and Week 12
  Questionnaires each consisting of 41 or fewer items on a Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Farias, PhD, Principal Investigator — University of California, Davis
Locations (1):
- Alzheimer's Disease Center, University of California, Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No
We are not planning to share individual participant data with other researchers.

REFERENCES:
- See also: Learn more or sign up for the study here! — https://studypages.com/s/the-digital-memory-notebook-training-to-improve-everyday-functioning-in-older-adults-with-mild-cognitive-impairment-518781/